CLINICAL TRIAL: NCT02880085
Title: Use of a Marker for Cartilage Damage to Differentiate the Diagnosis of Femural Acetabular Impingement From Extraarticular Pathologies.
Brief Title: Marker for FAI Diagnosis
Acronym: MarkerFAI
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Enrico Tassinari, Doctor, Istituto Ortopedico Rizzoli
Other Study IDs: 07/15
Record Dates: First submitted 2016-02-23; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Anesthetics, Local; Lidocaine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and urine samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Local anesthetic — local injection
  Other Names: Lidocaine

SUMMARY:
The diagnostic gold standard to differentiate FAI (femural acetabular impingement) from other muscular-tendinous pathologies is, actually, the injection of intra-articular anesthetic (lidocaine), with a pre- and post- evaluation of pain scale.

If, after injection, the pain disappears, the pain is probably due to an articular problem (FAI). This kind of differential diagnosis test has a sensibility of 100% and a specificity of 81%.

C-terminal telopeptide of type II collagen (CTXII) as cartilage degradation index, could be a marker, simply detectable, to assess the healthy of the cartilage status and could be measured in serum and urine.

DETAILED DESCRIPTION:
This study is observational-analytical and cross-sectional, because the same patient will receive both the diagnostic iter.

For the rules of Evidence-based Medicine (Brown et al., 2006), the definition of this study PICO is:

P (population)= all the patients with suspected FAI afferent to Orthopaedic-Traumatology and Prosthetic surgery and revisions of hip and knee implants

I (intervention)= enzyme-linked immunosorbent assay (ELISA) for C-terminal telopeptide of type II collagen (CTXII) in serum and urine

C (comparison)= intra-articular lidocaine injection

O (outcome)= sensibility/specificity of ELISA test

From a literature analysis the C-terminal telopeptide of type II collagen (CTXII) seem to be the best candidate for this kind of comparison. Some previous studies (Scarpellini et al, 2008) demonstrated that this marker could be used in this way, and, for this reason, the aim of this study is to investigate the sensibility and specificity of this marker in serum and urine, vs the actual diagnostic gold standard (anesthetic intra-articular injection).

If the marker will be equal or better than the actual gold standard, the clinical practice will have an improvement, because this kind of analysis is simply performing and less invasive for the patient.

The study will enroll 20 patients with suspected FAI between 18-45 years and of both the gender.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of suspected FAI
* Patients with clinical addressing to arthroscopy

Exclusion Criteria:

* Patients referring articular rheumatic pathologies
* Patients referring traumatic events in hip
* Patients wearing other hip prosthesis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 20 male and female, age range 18-45 recovered for suspicious FAI
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of partecipants with positive FAI by diagnostic gold standard (anesthetic injection) and negative response of FAI by dosing markers. | 1 year
  It will be valuated with ROCC curve of both the diagnostic protocols. The Diagnostic Gold standard (anesthetic injection) ascertains the presence of FAI when, after anesthetic injection, the measured pain considerably decreases or disappears, using tha VAS scale for pain. If the dosage of the markers will be higher of the assessed normal values in the cases of diagnosed FAI, with a higher or equal sensitivity and specificity (%), it will be demonstrated that this kind of diagnosis could be a good subtituite of the actual diagnostic gold standard (valuated with ROCC curve)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratorio Tecnologia Medica, Bologna, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly BT, Buly RL. Hip arthroscopy update. HSS J. 2005 Sep;1(1):40-8. doi: 10.1007/s11420-005-0105-3. PMID 18751808
- [Background] Mintz DN, Hooper T, Connell D, Buly R, Padgett DE, Potter HG. Magnetic resonance imaging of the hip: detection of labral and chondral abnormalities using noncontrast imaging. Arthroscopy. 2005 Apr;21(4):385-93. doi: 10.1016/j.arthro.2004.12.011. PMID 15800516
- [Background] Philippon MJ, Maxwell RB, Johnston TL, Schenker M, Briggs KK. Clinical presentation of femoroacetabular impingement. Knee Surg Sports Traumatol Arthrosc. 2007 Aug;15(8):1041-7. doi: 10.1007/s00167-007-0348-2. Epub 2007 May 12. PMID 17497126
- [Background] Burnett RS, Della Rocca GJ, Prather H, Curry M, Maloney WJ, Clohisy JC. Clinical presentation of patients with tears of the acetabular labrum. J Bone Joint Surg Am. 2006 Jul;88(7):1448-57. doi: 10.2106/JBJS.D.02806. PMID 16818969
- [Background] Simpson J, Sadri H, Villar R. Hip arthroscopy technique and complications. Orthop Traumatol Surg Res. 2010 Dec;96(8 Suppl):S68-76. doi: 10.1016/j.otsr.2010.09.010. Epub 2010 Oct 30. PMID 21036688